CLINICAL TRIAL: NCT00258154
Title: Safety and Immunogenicity of Concomitant Use of V260 and INFANRIX™ Hexa in Healthy Infants
Brief Title: V260 Study: Concomitant Use of V260 and INFANRIX™ Hexa in Healthy Infants (V260-010)
Status: Completed | Phase: Phase 3 | Type: Interventional
Sponsor: Merck Sharp & Dohme LLC (Industry)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: Double | Purpose: Treatment
Other Study IDs: V260-010; 2005_046
Record Dates: First submitted 2005-11-15; First posted 2005-11-24 (Estimated); Results first posted 2009-09-23 (Estimated); Last update posted 2015-10-06 (Estimated); Status verified 2015-10

CONDITIONS: Rotavirus Disease
MeSH Terms: conditions — Rotavirus Infections | interventions — Rotavirus Vaccines; Acetylglucosaminidase

STUDY DESIGN:
Who Masked: Participant, Investigator

ARMS (2):
- 1 (Experimental): RotaTeq/Infanrix Hexa
  Interventions: Biological: Rotavirus Vaccine, Live, Oral, Pentavalent; Biological: Comparator: Infanrix(tm) Hexa
- 2 (Placebo Comparator): Placebo/Infanrix Hexa
  Interventions: Biological: Comparator: placebo; Biological: Comparator: Infanrix(tm) Hexa

INTERVENTIONS:
Biological: Rotavirus Vaccine, Live, Oral, Pentavalent — 3 doses of rotavirus vaccine live, oral, pentavalent on Day 1, 28 to 42 days post dose 1 and 28 to 42 days post dose 2
  Arms: 1
Biological: Comparator: placebo — 3 doses of placebo to rotavirus vaccine live, oral, pentavalent on Day 1, 28 to 42 days post dose 1 and 28 to 42 days post dose 2
  Arms: 2
Biological: Comparator: Infanrix(tm) Hexa — 3 doses of oral Infanrix(tm) Hexa on Day 1, 28 to 42 days post dose 1 and 28 to 42 days post dose 2

SUMMARY:
The study is being conducted to demonstrate that the vaccine to prevent gastroenteritis due to rotavirus may be administered concomitantly with INFANRIX(tm)hexa without impairing the safety and immunogenicity of either vaccine.

ELIGIBILITY:
Inclusion Criteria:

* Healthy infant per investigator, 6 through 12 weeks of age

Exclusion Criteria:

* History of congenital abdominal disorders, intussusception, or abdominal surgery
* Known or suspected impairment of immunological function
* Known hypersensitivity to any component of the rotavirus vaccine
* Prior administration of any rotavirus vaccine
* Known hypersensitivity or contraindication to any component of INFANRIX(tm) hexa
* Any infant born from a known HBsAg-positive mother
* Prior administration of any oral polio vaccine
* Receipt of one or more doses of inactivated poliovirus vaccine, diptheria, tetanus and acellular pertussis vaccine, diptheria, tetanus and pertussis vaccine, Haemophilus influenzae type b vaccine, or any hepatitis B vaccine prior to the first vaccination, or receipt of any vaccines with these antigens at any time during the course of the study
* Fever, with a rectal temperature greater than or equal to 38.1 degree C (greater than or equal to 100.5 degree F) at the time of immunization
* History of known prior rotavirus gastroenteritis, chronic diarrhea, or failure to thrive
* Clinical evidence of active gastrointestinal illness
* Receipt of intramuscular, oral, or intravenous corticosteroid treatment within the 2 weeks prior to vaccination
* Infants residing in a household with an immunocompromised person
* Prior receipt of a blood transfusion or blood products
* Participation in another clinical study within 42 days before the beginning or anytime during the duration of the current clinical study
* Any infant who cannot be adequately followed for safety by a contact visit
* History of seizure disorders or prior history followed for safety by a contact visit
* Any condition that, in the opinion of the investigator, may interfere with the evaluation of the study objectives

Ages: 6 Weeks to 12 Weeks | Sex: All | Healthy Volunteers: Yes
Age Groups: Child
Enrollment: 403 (Actual)
Dates: Start 2006-02; Primary Completion 2006-11 (Actual); Study Completion 2006-11 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: Medical Monitor, Study Director — Merck Sharp & Dohme LLC

REFERENCES:
- [Result] Ciarlet M, He S, Lai S, Petrecz M, Yuan G, Liu GF, Mikviman E, Heaton PM, Panzer F, Rose T, Koller DY, Van Damme P, Schodel F. Concomitant use of the 3-dose oral pentavalent rotavirus vaccine with a 3-dose primary vaccination course of a diphtheria-tetanus-acellular pertussis-hepatitis B-inactivated polio-Haemophilus influenzae type b vaccine: immunogenicity and reactogenicity. Pediatr Infect Dis J. 2009 Mar;28(3):177-81. doi: 10.1097/INF.0b013e31818c0161. PMID 19209092

RESULTS

PARTICIPANT FLOW:
Recruitment Details: Enrollment occurred at 26 sites in Austria, Belgium, and Germany from 22Feb2006 (first subject in) to 13Nov2006 (last subject out). Cutoff date for all clinical and laboratory data from the Case Report Forms in-house was 08Jun2007. Access to the clinical database was granted on 15Jun2007.
Pre-assignment Details: Excluded from randomization were patients with history of congenital abdominal disorders, intussusception, or abdominal surgery; history of known prior rotavirus disease, chronic diarrhea, or failure to thrive, clinical evidence of active gastrointestinal illness and those with fever, a rectal temperature >38.1°C (>100.5°F) at time of immunization.
Groups:
- RotaTeq™ + INFANRIX Hexa: Subjects in Group 1 received 3 concomitant doses of RotaTeq™ and INFANRIX™ hexa ≥28 to ≤42 days apart.
- Placebo + INFANRIX Hexa: For subjects in Group 2, 3 concomitant doses of placebo were administered concomitantly with INFANRIX™ hexa at intervals of 4 to 6 weeks.
Period: Overall Study
Arm/Group | RotaTeq™ + INFANRIX Hexa | Placebo + INFANRIX Hexa
Started | 201 (Healthy infants who started in the RotaTeq™ concomitantly with INFANRIX™ hexa group.) | 202 (Healthy infants who started in the Placebo concomitantly with INFANRIX™ hexa group.)
Vaccinated at Visit 1 | 201 | 202
Vaccinated at Visit 2 | 198 | 198
Vaccinated at Visit 3 | 195 | 197
Completed | 192 (Subjects who completed the study.) | 195 (Subjects who completed the study.)
Not Completed | 9 | 7
Not completed — Adverse Event | 1 | 0
Not completed — Lost to Follow-up | 0 | 1
Not completed — Protocol Violation | 2 | 1
Not completed — Withdrawal by Subject | 3 | 4
Not completed — Patient Moved | 3 | 1

BASELINE CHARACTERISTICS:
Groups:
- Total: Total of all reporting groups
Arm/Group | RotaTeq™ + INFANRIX Hexa | Placebo + INFANRIX Hexa | Total
Number analyzed (Participants) | 201 | 202 | 403
Age, Customized [Number; unit: participants]
  5 Weeks of Age and Under | 1 | 0 | 1
  6-12 Weeks of Age | 199 | 202 | 401
  Over 12 Weeks of Age | 1 | 0 | 1
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 104 | 102 | 206
  Male | 97 | 100 | 197
Race/Ethnicity, Customized [Number; unit: Participants]
  Asian | 4 | 2 | 6
  Black | 10 | 11 | 21
  Multi-Racial | 1 | 2 | 3
  White | 186 | 187 | 373

OUTCOME MEASURES:

1. Primary Outcome: Immunogenicity of INFANRIX™ Hexa in Relation to Anti-hepatitis B Surface Antigen HBsAg, Predose 1
Description: Geometric Mean Titer (GMT)/antibody responses to RotaTeq™ and INFANRIX™ in relation to anti-hepatitis B surface antigen HBsAg at start of a 3-dose regimen
Time Frame: Day 1 of a 3-dose regimen
Population: All per-protocol subjects were included in the analysis of primary endpoints for polyribosylribitol phosphate (PRP) and hepatitis B surface antigen (HBsAg). Subjects listed in the Protocol Violation Memo were excluded from the immunogenicity analysis; N analyzed = number of subjects contributing to per protocol analysis.
Measure: Geometric Mean (95% Confidence Interval); unit: mIU/mL
Arm/Group | RotaTeq™ + INFANRIX Hexa | Placebo + INFANRIX Hexa
Number analyzed (Participants) | 185 | 184
mIU/mL | 12.7 [10.0 to 16.1] | 13.5 [10.5 to 17.4]

2. Secondary Outcome: Immunogenicity of INFANRIX™ Hexa in Relation to Serum Antibody Levels to Poliovirus Type 1 When Administered Concomitantly With RotaTeq™, Predose 1
Description: GMT of Poliovirus Type 1 in subjects with even allocation numbers, receiving RotaTeq™ + INFANRIX™ hexa compared to those receiving placebo + INFANRIX™ hexa at the start of a 3-dose regimen
Time Frame: Predose (Day 1 of a 3-dose regimen)
Population: Per Protocol Analysis on Subset A (subjects with even allocation numbers)
Measure: Geometric Mean (95% Confidence Interval); unit: Dilution Unit
Arm/Group | RotaTeq™ + INFANRIX Hexa | Placebo + INFANRIX Hexa
Number analyzed (Participants) | 97 | 67
Dilution Unit | 15.1 [11.3 to 20.2] | 18.3 [12.9 to 26.0]

3. Primary Outcome: Immunogenicity of INFANRIX™ Hexa in Relation to Anti-hepatitis B Surface Antigen HBsAg , at 42 Days After a 3-dose Regimen
Description: GMT/antibody responses to RotaTeq™ and INFANRIX™ in relation to anti-hepatitis B surface antigen HBsAg at 42 days after 3-dose regimen
Time Frame: 42 days after 3-dose regimen
Population: as for outcome 1
Measure: Geometric Mean (95% Confidence Interval); unit: mIU/mL
Arm/Group | RotaTeq™ + INFANRIX Hexa | Placebo + INFANRIX Hexa
Number analyzed (Participants) | 184 | 184
mIU/mL | 227.8 [189.2 to 274.2] | 261.0 [219.3 to 310.7]
Statistical Analysis 1: Comparison: RotaTeq™ + INFANRIX Hexa vs Placebo + INFANRIX Hexa; Test type: Non-Inferiority or Equivalence — non-inferiority criterion is that the lower limit of the 2-sided 95% confidence interval of the proportion difference (Rotateq+INFANRIX hexa group minus Placebo+INFANRIX hexa group) for subjects who achieve serum antibody levels of ≥ 10 mIU/mL greater than -10%; p < 0.001, Miettinen and Nurminen's; Comparing percentage difference with the non-inferiority margin of 10 percentage point with Miettinen and Nurminen's method; Percentage point difference = 0.0, 95% CI [-3.7 to 3.6] — Percentage point difference (RotaTeq - Placebo)

4. Primary Outcome: Immunogenicity of INFANRIX™ Hexa in Relation to Serum Anti-polyribosylribitol Phosphate PRP, Predose 1
Description: GMT/antibody responses to RotaTeq™ and INFANRIX™ hexa in relation to serum anti-polyribosylribitol phosphate PRP at start of 3-dose regimen
Time Frame: Day 1 of 3-dose regimen
Population: as for outcome 1
Measure: Geometric Mean (95% Confidence Interval); unit: ng/mL
Arm/Group | RotaTeq™ + INFANRIX Hexa | Placebo + INFANRIX Hexa
Number analyzed (Participants) | 184 | 184
ng/mL | 204.3 [181.6 to 229.8] | 189.7 [170.0 to 211.8]

5. Primary Outcome: Immunogenicity of INFANRIX™ Hexa in Relation to Serum Anti-polyribosylribitol Phosphate PRP at 42 Days After a 3-dose Regimen
Description: GMT/antibody responses to RotaTeq™ and INFANRIX™ hexa in relation to serum anti-polyribosylribitol phosphate PRP at 42 days after a 3-dose regimen
Time Frame: 42 days after a 3-dose regimen
Population: as for outcome 1
Measure: Geometric Mean (95% Confidence Interval); unit: ng/mL
Arm/Group | RotaTeq™ + INFANRIX Hexa | Placebo + INFANRIX Hexa
Number analyzed (Participants) | 185 | 184
ng/mL | 1316 [1081 to 1603] | 1400 [1172 to 1672]
Statistical Analysis 1: Comparison: RotaTeq™ + INFANRIX Hexa vs Placebo + INFANRIX Hexa; Test type: Non-Inferiority or Equivalence — non-inferiority criterion is that the lower limit of the 2-sided 95% confidence interval of the proportion difference (Rotateq+INFANRIX hexa group minus Placebo+INFANRIX hexa group) for subjects who achieve serum antibody levels of ≥ 0.15 μg/mL greater than -10%; p = 0.015, Miettinen and Nurminen's; [statistical method as in outcome 3, analysis 1]; Percentage point difference = -3.7, 95% CI [-9.3 to 1.3] — Percentage point difference (RotaTeq - Placebo)

6. Secondary Outcome: Immunogenicity of INFANRIX™ Hexa in Relation to Serum Antibody Levels to Poliovirus Type 1 When Administered Concomitantly With RotaTeq™, 42 Days After a 3-dose Regimen
Description: GMT of Poliovirus Type 1 in subjects with even allocation numbers, receiving RotaTeq™ + INFANRIX™ hexa compared to those receiving placebo + INFANRIX™ hexa , 42 days after a 3-dose regimen
Time Frame: 42 days after a 3-dose regimen
Population: Per Protocol Analysis on Subset A (subjects with even allocation numbers)
Measure: Geometric Mean (95% Confidence Interval); unit: Dilution Unit
Arm/Group | RotaTeq™ + INFANRIX Hexa | Placebo + INFANRIX Hexa
Number analyzed (Participants) | 95 | 68
Dilution Unit | 94.9 [68.9 to 130.6] | 160.2 [113.6 to 225.8]

7. Secondary Outcome: Immunogenicity of INFANRIX™ Hexa in Relation to Serum Antibody Levels to Poliovirus Type 2 When Administered Concomitantly With RotaTeq™, Predose 1
Description: GMT of Poliovirus Type 2 in subjects with even allocation numbers, receiving RotaTeq™ + INFANRIX™ hexa compared to those receiving placebo + INFANRIX™ hexa at the start of a 3-dose regimen
Time Frame: Pre-dose (Day 1 of a 3-dose regimen)
Population: Per Protocol Analysis on Subset A (subjects with even allocation numbers)
Measure: Geometric Mean (95% Confidence Interval); unit: Dilution Unit
Arm/Group | RotaTeq™ + INFANRIX Hexa | Placebo + INFANRIX Hexa
Number analyzed (Participants) | 97 | 67
Dilution Unit | 12.8 [9.8 to 16.8] | 12.7 [9.2 to 17.6]

8. Secondary Outcome: Immunogenicity of INFANRIX™ Hexa in Relation to Serum Antibody Levels to Poliovirus Type 2 When Administered Concomitantly With RotaTeq™, 42 Days After a 3-dose Regimen
Description: GMT of Poliovirus Type 2 in subjects with even allocation numbers, receiving RotaTeq™ + INFANRIX™ hexa compared to those receiving placebo + INFANRIX™ hexa 42 days after a 3-dose regimen
Time Frame: 42 days after in a 3-dose regimen
Population: Per Protocol Analysis on Subset A (subjects with even allocation numbers)
Measure: Geometric Mean (95% Confidence Interval); unit: Dilution Unit
Arm/Group | RotaTeq™ + INFANRIX Hexa | Placebo + INFANRIX Hexa
Number analyzed (Participants) | 95 | 68
Dilution Unit | 63.1 [45.8 to 86.8] | 69.4 [48.6 to 99.2]

9. Secondary Outcome: Immunogenicity of INFANRIX™ Hexa in Relation to Serum Antibody Levels to Poliovirus Type 3 When Administered Concomitantly With RotaTeq™, Predose 1
Description: GMT of Poliovirus Type 3 in subjects with even allocation numbers, receiving RotaTeq™ + INFANRIX™ hexa compared to those receiving placebo + INFANRIX™ hexa at the start of a 3-dose regimen
Time Frame: Predose (Day 1 of a 3-dose regimen)
Population: Per Protocol Analysis on Subset A (subjects with even allocation numbers)
Measure: Geometric Mean (95% Confidence Interval); unit: Dilution Unit
Arm/Group | RotaTeq™ + INFANRIX Hexa | Placebo + INFANRIX Hexa
Number analyzed (Participants) | 97 | 67
Dilution Unit | 9.0 [6.8 to 12.1] | 7.8 [5.7 to 10.7]

10. Secondary Outcome: Immunogenicity of INFANRIX™ Hexa in Relation to Serum Antibody Levels to Poliovirus Type 3 When Administered Concomitantly With RotaTeq™, 42 Days After a 3-dose Regimen
Description: GMT of Poliovirus Type 3 in subjects with even allocation numbers, receiving RotaTeq™ + INFANRIX™ hexa compared to those receiving placebo + INFANRIX™ hexa 42 days after a 3-dose regimen
Time Frame: 42 days after a 3-dose regimen
Population: Per Protocol Analysis on Subset A (subjects with even allocation numbers)
Measure: Geometric Mean (95% Confidence Interval); unit: Dilution Unit
Arm/Group | RotaTeq™ + INFANRIX Hexa | Placebo + INFANRIX Hexa
Number analyzed (Participants) | 95 | 68
Dilution Unit | 222.9 [153.9 to 322.8] | 263.9 [173.5 to 401.5]

11. Secondary Outcome: Immunogenicity of INFANRIX™ Hexa in Relation to Serum Antibody Levels to Diphtheria Toxoid When Administered Concomitantly With RotaTeq™, Predose 1
Description: GMT of diphtheria toxoid in subjects with odd allocation numbers, receiving RotaTeq™ + INFANRIX™ hexa compared to those receiving placebo + INFANRIX™ hexa at the start of a 3-dose regimen
Time Frame: Predose (Day 1 of a 3-dose regimen)
Population: Per Protocol Analysis on Subset B (subjects with odd allocation number)
Measure: Geometric Mean (95% Confidence Interval); unit: IU/mL
Arm/Group | RotaTeq™ + INFANRIX Hexa | Placebo + INFANRIX Hexa
Number analyzed (Participants) | 78 | 104
IU/mL | 0.0 [0.0 to 0.0] | 0.0 [0.0 to 0.1]

12. Secondary Outcome: Immunogenicity of INFANRIX™ Hexa in Relation to Serum Antibody Levels to Diphtheria Toxoid When Administered Concomitantly With RotaTeq™, 42 Days After a 3-dose Regimen
Description: GMT of diphtheria toxoid in subjects with odd allocation numbers, receiving RotaTeq™ + INFANRIX™ hexa compared to those receiving placebo + INFANRIX™ hexa 42 days after a 3-dose regimen
Time Frame: 42 days after a 3-dose regimen
Population: Per Protocol Analysis on Subset B (subjects with odd allocation number)
Measure: Geometric Mean (95% Confidence Interval); unit: IU/mL
Arm/Group | RotaTeq™ + INFANRIX Hexa | Placebo + INFANRIX Hexa
Number analyzed (Participants) | 73 | 100
IU/mL | 0.1 [0.1 to 0.1] | 0.1 [0.1 to 0.1]

13. Secondary Outcome: Immunogenicity of INFANRIX™ Hexa in Relation to Serum Antibody Levels to Tetanus Toxoid When Administered Concomitantly With RotaTeq™, Predose 1
Description: GMT of tetanus toxoid in subjects with odd allocation numbers, receiving RotaTeq™ + INFANRIX™ hexa compared to those receiving placebo + INFANRIX™ hexa at the start of a 3-dose regimen
Time Frame: Predose (Day 1 of a 3-dose regimen)
Population: Per Protocol Analysis on Subset B (subjects with odd allocation numbers)
Measure: Geometric Mean (95% Confidence Interval); unit: IU/mL
Arm/Group | RotaTeq™ + INFANRIX Hexa | Placebo + INFANRIX Hexa
Number analyzed (Participants) | 76 | 104
IU/mL | 0.2 [0.2 to 0.4] | 0.3 [0.2 to 0.5]

14. Secondary Outcome: Immunogenicity of INFANRIX™ Hexa in Relation to Serum Antibody Levels to Tetanus Toxoid When Administered Concomitantly With RotaTeq™, 42 Days After a 3-dose Regimen
Description: GMT of tetanus toxoid in subjects with odd allocation numbers, receiving RotaTeq™ + INFANRIX™ hexa compared to those receiving placebo + INFANRIX™ hexa 42 days after a 3-dose regimen
Time Frame: 42 days after a 3-dose regimen
Population: Per Protocol Analysis on Subset B (subjects with odd allocation numbers
Measure: Geometric Mean (95% Confidence Interval); unit: Dilution Unit
Arm/Group | RotaTeq™ + INFANRIX Hexa | Placebo + INFANRIX Hexa
Number analyzed (Participants) | 72 | 101
Dilution Unit | 1.4 [1.1 to 1.7] | 1.5 [1.2 to 1.8]

15. Secondary Outcome: Immunogenicity of INFANRIX™ Hexa in Relation to Serum Antibody Levels to Pertussis FHA When Administered Concomitantly With RotaTeq™, Predose 1
Description: GMT of pertussis FHA in subjects receiving RotaTeq™ + INFANRIX™ hexa compared to those receiving placebo + INFANRIX™ hexa at the start of a 3-dose regimen
Time Frame: Predose (Day 1 of a 3-dose regimen)
Population: Per Protocol Analysis
Measure: Geometric Mean (95% Confidence Interval); unit: EU/mL
Arm/Group | RotaTeq™ + INFANRIX Hexa | Placebo + INFANRIX Hexa
Number analyzed (Participants) | 180 | 177
EU/mL | 4.3 [3.2 to 5.9] | 3.7 [2.7 to 5.1]

16. Secondary Outcome: Immunogenicity of INFANRIX™ Hexa in Relation to Serum Antibody Levels to Pertussis FHA When Administered Concomitantly With RotaTeq™, 42 Days After a 3-dose Regimen
Description: GMT of pertussis FHA in subjects receiving RotaTeq™ + INFANRIX™ hexa compared to those receiving placebo + INFANRIX™ hexa 42 days after a 3-dose regimen
Time Frame: 42 days after a 3-dose regimen
Population: Per Protocol Analysis
Measure: Least Squares Mean (95% Confidence Interval); unit: EU/mL
Arm/Group | RotaTeq™ + INFANRIX Hexa | Placebo + INFANRIX Hexa
Number analyzed (Participants) | 177 | 176
EU/mL | 74 [67.2 to 81.4] | 78.8 [71.6 to 86.7]

17. Secondary Outcome: Immunogenicity of INFANRIX™ Hexa in Relation to Serum Antibody Levels to Pertussis Pertactin When Administered Concomitantly With RotaTeq™, Predose 1
Description: GMT of pertussis Pertactin in subjects receiving RotaTeq™ + INFANRIX™ hexa compared to those receiving placebo + INFANRIX™ hexa at the start of a 3-dose regimen
Time Frame: Predose (Day 1 of a 3-dose regimen)
Population: Per Protocol Analysis
Measure: Geometric Mean (95% Confidence Interval); unit: EU/mL
Arm/Group | RotaTeq™ + INFANRIX Hexa | Placebo + INFANRIX Hexa
Number analyzed (Participants) | 180 | 177
EU/mL | 1.0 [0.7 to 1.4] | 1.0 [0.7 to 1.4]

18. Secondary Outcome: Immunogenicity of INFANRIX™ Hexa in Relation to Serum Antibody Levels to Pertussis Pertactin When Administered Concomitantly With RotaTeq™, 42 Days After a 3-dose Regimen
Description: GMT of pertussis Pertactin in subjects receiving RotaTeq™ + INFANRIX™ hexa compared to those receiving placebo + INFANRIX™ hexa 42 days after a 3-dose regimen
Time Frame: 42 days after a 3-dose regimen
Population: Per Protocol Analysis
Measure: Geometric Mean (95% Confidence Interval); unit: EU/mL
Arm/Group | RotaTeq™ + INFANRIX Hexa | Placebo + INFANRIX Hexa
Number analyzed (Participants) | 177 | 177
EU/mL | 109.6 [96.7 to 124.1] | 108.2 [93.5 to 125.1]

19. Secondary Outcome: Immunogenicity of INFANRIX™ Hexa in Relation to Serum Antibody Levels to Pertussis Toxoid When Administered Concomitantly With RotaTeq™, Predose 1
Description: GMT of pertussis toxoid in subjects receiving RotaTeq™ + INFANRIX™ hexa compared to those receiving placebo + INFANRIX™ hexa at the start of a 3-dose regimen
Time Frame: Predose (Day 1 of a 3-dose regimen)
Population: Per Protocol Analysis
Measure: Geometric Mean (95% Confidence Interval); unit: EU/mL
Arm/Group | RotaTeq™ + INFANRIX Hexa | Placebo + INFANRIX Hexa
Number analyzed (Participants) | 180 | 177
EU/mL | 0.2 [0.2 to 0.2] | 0.2 [0.2 to 0.3]

20. Secondary Outcome: Immunogenicity of INFANRIX™ Hexa in Relation to Serum Antibody Levels to Pertussis Toxoid When Administered Concomitantly With RotaTeq™, 42 Days After a 3-dose Regimen
Description: GMT of pertussis toxoid in subjects receiving RotaTeq™ + INFANRIX™ hexa compared to those receiving placebo + INFANRIX™ hexa 42 days after a 3-dose regimen
Time Frame: 42 days after a 3-dose regimen
Population: Per Protocol Analysis
Measure: Geometric Mean (95% Confidence Interval); unit: EU/mL
Arm/Group | RotaTeq™ + INFANRIX Hexa | Placebo + INFANRIX Hexa
Number analyzed (Participants) | 177 | 176
EU/mL | 28.0 [24.8 to 31.7] | 28.3 [25.2 to 31.8]

21. Secondary Outcome: Serum Neutralizing Antibody (SNA) Response to Serotype G1 in Patients Receiving RotaTeq™ Concomitantly With INFANRIX™ Hexa, Predose 1
Description: GMT of serotype G1 in subjects receiving RotaTeq™ + INFANRIX™ hexa compared to those receiving placebo + INFANRIX™ hexa at the start of a 3-dose regimen
Time Frame: Predose (Day 1 of a 3-dose regimen)
Population: Per Protocol Analysis
Measure: Geometric Mean (95% Confidence Interval); unit: GMT
Arm/Group | RotaTeq™ + INFANRIX Hexa | Placebo + INFANRIX Hexa
Number analyzed (Participants) | 184 | 182
GMT | 23.3 [19.6 to 27.7] | 24 [20.3 to 28.4]

22. Secondary Outcome: Serum Neutralizing Antibody (SNA) Response to Serotype G1 in Patients Receiving RotaTeq™ Concomitantly With INFANRIX™ Hexa, 42 Days After a 3-dose Regimen
Description: GMT of serotype G1 in subjects receiving RotaTeq™ + INFANRIX™ hexa compared to those receiving placebo + INFANRIX™ hexa 42 days after a 3-dose regimen
Time Frame: 42 days after a 3-dose regimen
Population: Per Protocol Analysis
Measure: Geometric Mean (95% Confidence Interval); unit: GMT
Arm/Group | RotaTeq™ + INFANRIX Hexa | Placebo + INFANRIX Hexa
Number analyzed (Participants) | 184 | 183
GMT | 115.7 [94.2 to 142.1] | 8.2 [7.2 to 9.3]

23. Secondary Outcome: Serum Neutralizing Antibody (SNA) Response to Serotype G2 in Patients Receiving RotaTeq™ Concomitantly With INFANRIX™ Hexa, Predose 1
Description: GMT of serotype G2 in subjects receiving RotaTeq™ + INFANRIX™ hexa compared to those receiving placebo + INFANRIX™ hexa at the start of a 3-dose regimen
Time Frame: Predose (Day 1 of a 3-dose regimen)
Population: Per Protocol Analysis
Measure: Geometric Mean (95% Confidence Interval); unit: GMT
Arm/Group | RotaTeq™ + INFANRIX Hexa | Placebo + INFANRIX Hexa
Number analyzed (Participants) | 184 | 181
GMT | 11.7 [10.2 to 13.4] | 12.2 [10.6 to 14.1]

24. Secondary Outcome: Serum Neutralizing Antibody (SNA) Response to Serotype G2 in Patients Receiving RotaTeq™ Concomitantly With INFANRIX™ Hexa 42 Days After a 3-dose Regimen
Description: GMT of serotype G2 in subjects receiving RotaTeq™ + INFANRIX™ hexa compared to those receiving placebo + INFANRIX™ hexa 42 days after a 3-dose regimen
Time Frame: 42 days after a 3-dose regimen
Population: Per Protocol Analysis
Measure: Geometric Mean (95% Confidence Interval); unit: GMT
Arm/Group | RotaTeq™ + INFANRIX Hexa | Placebo + INFANRIX Hexa
Number analyzed (Participants) | 184 | 183
GMT | 16.6 [14.0 to 19.7] | 6.1 [5.6 to 6.6]

25. Secondary Outcome: Serum Neutralizing Antibody (SNA) Response to Serotype G3 in Patients Receiving RotaTeq™ Concomitantly With INFANRIX™ Hexa Predose 1
Description: GMT of serotype G3 in subjects receiving RotaTeq™ + INFANRIX™ hexa compared to those receiving placebo + INFANRIX™ hexa Predose 1
Time Frame: Predose (Day 1 of a 3-dose regimen)
Population: Per Protocol Analysis
Measure: Geometric Mean (95% Confidence Interval); unit: GMT
Arm/Group | RotaTeq™ + INFANRIX Hexa | Placebo + INFANRIX Hexa
Number analyzed (Participants) | 184 | 182
GMT | 11.5 [9.7 to 13.6] | 9.8 [8.5 to 11.3]

26. Secondary Outcome: Serum Neutralizing Antibody (SNA) Response to Serotype G3 in Patients Receiving RotaTeq™ Concomitantly With INFANRIX™ Hexa 42 Days After a 3-dose Regimen
Description: GMT of serotype G3 in subjects receiving RotaTeq™ + INFANRIX™ hexa compared to those receiving placebo + INFANRIX™ hexa 42 days after a 3-dose regimen
Time Frame: 42 days after a 3-dose regimen
Population: Per Protocol Analysis
Measure: Geometric Mean (95% Confidence Interval); unit: GMT
Arm/Group | RotaTeq™ + INFANRIX Hexa | Placebo + INFANRIX Hexa
Number analyzed (Participants) | 184 | 183
GMT | 28.0 [23.4 to 33.5] | 5.8 [5.5 to 6.3]

27. Secondary Outcome: Serum Neutralizing Antibody (SNA) Response to Serotype G4 in Patients Receiving RotaTeq™ Concomitantly With INFANRIX™ Hexa Predose 1
Description: GMT of serotype G4 in subjects receiving RotaTeq™ + INFANRIX™ hexa compared to those receiving placebo + INFANRIX™ hexa Predose 1
Time Frame: Predose (Day 1 of a 3-dose regimen)
Population: Per Protocol Analysis
Measure: Geometric Mean (95% Confidence Interval); unit: GMT
Arm/Group | RotaTeq™ + INFANRIX Hexa | Placebo + INFANRIX Hexa
Number analyzed (Participants) | 184 | 182
GMT | 15.5 [12.9 to 18.6] | 17.9 [15.0 to 21.3]

28. Secondary Outcome: Serum Neutralizing Antibody (SNA) Response to Serotype G4 in Patients Receiving RotaTeq™ Concomitantly With INFANRIX™ Hexa 42 Days After a 3-dose Regimen
Description: GMT of serotype G4 in subjects receiving RotaTeq™ + INFANRIX™ hexa compared to those receiving placebo + INFANRIX™ hexa 42 days after a 3-dose regimen
Time Frame: 42 days after a 3-dose regimen
Population: Per Protocol Analysis
Measure: Geometric Mean (95% Confidence Interval); unit: GMT
Arm/Group | RotaTeq™ + INFANRIX Hexa | Placebo + INFANRIX Hexa
Number analyzed (Participants) | 184 | 183
GMT | 33.6 [28.6 to 39.6] | 7.1 [6.5 to 7.7]

29. Secondary Outcome: Serum Neutralizing Antibody (SNA) Response to Serotype P1A in Patients Receiving RotaTeq™ Concomitantly With INFANRIX™ Hexa Predose 1
Description: GMT of serotype P1A in subjects receiving RotaTeq™ + INFANRIX™ hexa compared to those receiving placebo + INFANRIX™ hexa Predose 1
Time Frame: Predose (Day 1 of a 3-dose regimen)
Population: Per Protocol Analysis
Measure: Geometric Mean (95% Confidence Interval); unit: GMT
Arm/Group | RotaTeq™ + INFANRIX Hexa | Placebo + INFANRIX Hexa
Number analyzed (Participants) | 184 | 181
GMT | 36.8 [30.9 to 44.0] | 33.2 [28.1 to 39.3]

30. Secondary Outcome: Serum Neutralizing Antibody (SNA) Response to Serotype P1A in Patients Receiving RotaTeq™ Concomitantly With INFANRIX™ Hexa 42 Days After a 3-dose Regimen
Description: GMT of serotype P1A in subjects receiving RotaTeq™ + INFANRIX™ hexa compared to those receiving placebo + INFANRIX™ hexa 42 days after a 3-dose regimen
Time Frame: 42 days after a 3-dose regimen
Population: Per Protocol Analysis
Measure: Geometric Mean (95% Confidence Interval); unit: GMT
Arm/Group | RotaTeq™ + INFANRIX Hexa | Placebo + INFANRIX Hexa
Number analyzed (Participants) | 184 | 183
GMT | 74.5 [60.7 to 91.3] | 10.7 [9.2 to 12.4]

31. Secondary Outcome: Serum Neutralizing Antibody (SNA) Response to Serum Anti-rotavirus IgA in Patients Receiving RotaTeq™ Concomitantly With INFANRIX™ Hexa Predose 1
Description: GMT of serum anti-rotavirus IgA in subjects receiving RotaTeq™ + INFANRIX™ hexa compared to those receiving placebo + INFANRIX™ hexa Predose 1
Time Frame: Predose (Day 1 of a 3-dose regimen)
Population: Per Protocol Analysis
Measure: Geometric Mean (95% Confidence Interval); unit: GMT
Arm/Group | RotaTeq™ + INFANRIX Hexa | Placebo + INFANRIX Hexa
Number analyzed (Participants) | 184 | 181
GMT | 0.1 [0.1 to 0.2] | 0.1 [0.1 to 0.2]

32. Secondary Outcome: Serum Neutralizing Antibody (SNA) Response to Serum Anti-rotavirus IgA in Patients Receiving RotaTeq™ Concomitantly With INFANRIX™ Hexa 42 Days After a 3-dose Regimen
Description: GMT of serum anti-rotavirus IgA in subjects receiving RotaTeq™ + INFANRIX™ hexa compared to those receiving placebo + INFANRIX™ hexa 42 days after a 3-dose regimen
Time Frame: 42 days after a 3-dose regimen
Population: Per Protocol Analysis
Measure: Geometric Mean (95% Confidence Interval); unit: GMT
Arm/Group | RotaTeq™ + INFANRIX Hexa | Placebo + INFANRIX Hexa
Number analyzed (Participants) | 184 | 183
GMT | 160.0 [119.0 to 215.3] | 0.2 [0.1 to 0.2]

ADVERSE EVENTS:
Time Frame: Patients in this study were followed for all adverse experiences, for 14 days following each study vaccination.
Description: The number of patients listed in the Adverse Event tables is the number of patients who received study treatment.
  Although a patient may have had two or more clinical adverse experiences the patient is counted only once in a category. The same patient may appear in different categories.
Arm/Group | RotaTeq™ + INFANRIX Hexa | Placebo + INFANRIX Hexa
Serious Adverse Events (participants affected / at risk) | 3/201 | 6/202
Other Adverse Events (participants affected / at risk) | 166/201 | 167/202
SERIOUS ADVERSE EVENTS; cells are participants affected of the arm's N at risk:
Term (organ system) | RotaTeq™ + INFANRIX Hexa (N=201) | Placebo + INFANRIX Hexa (N=202)
Abdominal symptom (Gastrointestinal disorders) | 0 | 1
Enteritis (Gastrointestinal disorders) | 0 | 1
Vomiting (Gastrointestinal disorders) | 0 | 1
Pyrexia (General disorders) | 0 | 2
Gastroenteritis salmonella (Infections and infestations) | 0 | 1
Pyelonephritis (Infections and infestations) | 0 | 1
Accidental overdose (Injury, poisoning and procedural complications) | 1 | 1
Concussion (Injury, poisoning and procedural complications) | 1 | 1
Head injury (Injury, poisoning and procedural complications) | 1 | 0
Dehydration (Metabolism and nutrition disorders) | 0 | 1
Crying (Psychiatric disorders) | 0 | 1
Restlessness (Psychiatric disorders) | 0 | 1
OTHER ADVERSE EVENTS (reported when occurring in more than 2% of participants in an arm); cells are participants affected of the arm's N at risk:
Term (organ system) | RotaTeq™ + INFANRIX Hexa (N=201) | Placebo + INFANRIX Hexa (N=202)
Conjunctivitis (Eye disorders) | 8 | 3
Abdominal pain (Gastrointestinal disorders) | 8 | 8
Diarrhoea (Gastrointestinal disorders) | 57 | 65
Enteritis (Gastrointestinal disorders) | 27 | 28
Flatulence (Gastrointestinal disorders) | 9 | 5
Vomiting (Gastrointestinal disorders) | 62 | 48
Irritability (General disorders) | 7 | 4
Pain (General disorders) | 4 | 2
Pyrexia (General disorders) | 106 | 114
Nasopharyngitis (Infections and infestations) | 8 | 6
Oral candidiasis (Infections and infestations) | 3 | 5
Respiratory tract infection (Infections and infestations) | 4 | 3
Rhinitis (Infections and infestations) | 11 | 17
Upper respiratory tract infection (Infections and infestations) | 2 | 5
Viral infection (Infections and infestations) | 5 | 2
Somnolence (Nervous system disorders) | 7 | 4
Crying (Psychiatric disorders) | 6 | 7
Restlessness (Psychiatric disorders) | 11 | 16
Cough (Respiratory, thoracic and mediastinal disorders) | 8 | 11
Rash (Skin and subcutaneous tissue disorders) | 4 | 1

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: No; Agreement restricts PI disclosure of results: Yes; Restriction type: Other
Merck agreements may vary with individual investigators, but will not prohibit any investigator from publishing. Merck supports the publication of results from all centers of a multi-center trial but requests that reports based on single-site data not precede the primary publication of the entire clinical trial.